CLINICAL TRIAL: NCT02519166
Title: Characterisation of Biofilm of the Chronic Wounds
Acronym: Biofilm Plaie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2012-02
Record Dates: First submitted 2015-07-28; First posted 2015-08-10 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Chronic Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with chronic wounds (Other)
  Interventions: Biological: 1 clinical examination of the wound, 1 sample taken with the curette, 1 sample by swabbing

INTERVENTIONS:
Biological: 1 clinical examination of the wound, 1 sample taken with the curette, 1 sample by swabbing

SUMMARY:
In this prospective observational study, the investigators tried assess the presence of biofilm on chronic wound samples coming from a large cohort study of patients, whilst cross-referencing the clinical, bacteriological and wound care observations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic wounds (period > 6 weeks) > 10 cm2
* Patient age >18 for the 3 French centres
* Patient participation in a follow-up program for treatment of their wound > 1 month
* Availability of patient information and written informed consent from them or their legal representative

Exclusion Criteria:

* Patients unable to submit to medical follow-up in the trial due to geographical constraints etc
* Patients deprived of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical examination | 1 month
characterisation of biofilm by fluorescence microscopy and confocal | 1 month

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Chu Montpellier, Montpellier
  - Institut Curie, Paris
  - Hopital Rothschild, Paris